CLINICAL TRIAL: NCT00012597
Title: Pressure Ulcer Assessment Via Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACC 97-013
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Web-based telemedicine system for assessment of status of pressure ulcers

INTERVENTIONS:
Procedure: Web-based telemedicine system for assessment of status of pressure ulcers

SUMMARY:
A Web-based telemedicine system for monitoring the status of patients with pressure ulcers has been developed. It consists of three major data collection components: (1) digital photograph of ulcer; (2) quantitative measurements of wound status (i.e., ulcer area and volume, skin elasticity); and (3) other wound and patient data collected by a nurse. Data are collected via laptop computer and transmitted to a central database, where a computer program transforms the data into the necessary reporting format. The output is posted onto a World Wide Web page for access by the consulting physician. The system incorporates all data requirements for assessment recommended by AHCPR's Clinical Practice Guideline, Treatment of Pressure Ulcers.

DETAILED DESCRIPTION:
Background:

A Web-based telemedicine system for monitoring the status of patients with pressure ulcers has been developed. It consists of three major data collection components: (1) digital photograph of ulcer; (2) quantitative measurements of wound status (i.e., ulcer area and volume, skin elasticity); and (3) other wound and patient data collected by a nurse. Data are collected via laptop computer and transmitted to a central database, where a computer program transforms the data into the necessary reporting format. The output is posted onto a World Wide Web page for access by the consulting physician. The system incorporates all data requirements for assessment recommended by AHCPR's Clinical Practice Guideline, Treatment of Pressure Ulcers.

Objectives:

The primary objective of this pilot study was to evaluate the clinical accuracy of a telemedicine system for assessing the status of pressure ulcers, both chronic and those which have been surgically repaired. The principal hypotheses were: (1) use of the telemedicine system results in the same diagnoses as does in-person patient assessment; and (2) patients are satisfied with the telemedicine system.

Methods:

Two VA medical centers and two specialties participated in the study: Ann Arbor (plastic surgery) and Augusta (plastic surgery, physical medicine and rehabilitation). They contributed inpatients and outpatients with a pressure ulcer of stage II, III, or IV over a one-year enrollment period. All study patients were assessed both in-person (the "gold standard") and with the telemedicine system. The in-person and telemedicine physicians provided yes/no responses to four diagnostic questions concerning wound healing and infection, based on AHCPR guidelines, and they were blinded to each other�s assessments. Patient satisfaction data were collected using a specially designed, self-administered questionnaire to measure perceptions regarding the burden of the telemedicine system, confidence in the evaluation, and absence of direct contact with a physician.

Status:

Completed

ELIGIBILITY:
Inclusion Criteria:

VA inpatients, outpatients, or nursing home residents at the participating sites who have any of the following wounds: (1) chronic pressure ulcers at stage II, III or IV; (2) post-operative wound patients having undergone a skin flap procedure for a grade III or IV pressure ulcer; (3) diabetic wounds; (4) arterial ulcers; or (5) chronic venous status ulcers. Exclusion criteria: Mentally incompetent patients.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie C Lowery, PhD MHSA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan

REFERENCES:
- [Result] Kim HM, Lowery JC, Hamill JB, Wilkins EG. Accuracy of a web-based system for monitoring chronic wounds. Telemed J E Health. 2003 Summer;9(2):129-40. doi: 10.1089/153056203766437471. PMID 12855036
- [Result] Kim HM, Lowery JC, Hamill JB, Wilkins EG. Patient attitudes toward a Web-based system for monitoring chronic wounds. Telemed J E Health. 2004;10 Suppl 2:S-26-34. PMID 23570210
- [Result] Lowery JC, Hamill JB, Wilkins EG, Clements E. Technical overview of a web-based telemedicine system for wound assessment. Adv Skin Wound Care. 2002 Jul-Aug;15(4):165-6, 168-9. doi: 10.1097/00129334-200207000-00007. PMID 12151982
- [Result] Roth RS, Lowery JC, Hamill JB. Assessing persistent pain and its relation to affective distress, depressive symptoms, and pain catastrophizing in patients with chronic wounds: a pilot study. Am J Phys Med Rehabil. 2004 Nov;83(11):827-34. doi: 10.1097/01.phm.0000140800.83146.fa. PMID 15502735
- [Result] Wilkins EG, Lowery JC, Goldfarb S. Feasibility of virtual wound care: a pilot study. Adv Skin Wound Care. 2007 May;20(5):275-6, 278. doi: 10.1097/01.ASW.0000269315.30639.82. PMID 17473564